CLINICAL TRIAL: NCT02795754
Title: A Double-Blind (Sponsor Unblinded), Randomized, Placebo-Controlled, Continuation Single and Repeated Dose Escalation Study to Investigate the Safety, Tolerability and Pharmacokinetics of GSK2838232 With Ritonavir, in Healthy Subjects
Brief Title: Single and Repeated Dose Escalation Study of GSK2838232
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 204953
Record Dates: First submitted 2016-01-21; First posted 2016-06-10 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: GSK2838232; HIV; repeated dose escalation; immediate release tablet; single dose escalation
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — Ritonavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- GSK2838232 PIB (50 mg+100 mg+200 mg)+Placebo (Experimental): During Part 1A, subjects will receive QD single dose of either GSK2838232 50 mg, 100 mg or 200 mg or placebo in each of the four visits (one treatment per visit).Subjects will also receive RTV along with all the doses and QD RTV for 48hours (2 doses) before all doses of GSK2838232 and placebo.
  Interventions: Drug: GSK2838232 PIB; Drug: Placebo PIB; Drug: Ritonavir
- GSK2838232 PIB+IR1+IR2 (Experimental): During Part 1B, subjects will receive either GSK2838232 PIB, GSK2838232 IR1 or IR2 in each of the three visits (one treatment per visit) after at least 10 hours fasting and IR1 or IR2 after fat meal at visit 4.
  Interventions: Drug: GSK2838232 PIB; Drug: GSK2838232 IR1; Drug: GSK2838232 IR2; Drug: Ritonavir
- GSK2838232 PIB (20mg/50 mg/100 mg/200 mg)/Placebo (Experimental): During Part 2, subjects will receive repeated QD doses of either GSK2838232 (20 mg, 50 mg, 100 mg or 200 mg) or placebo for 11 days. Subjects will also receive RTV along with all the doses of GSK2838232 and placebo.
  Interventions: Drug: GSK2838232 PIB; Drug: Placebo PIB; Drug: Ritonavir

INTERVENTIONS:
Drug: GSK2838232 PIB — GSK2838232 will be available as oral suspension for reconstitution, will be administered as 50, 100 and 200 mg in Part A and as 20, 50, 100 or 200 mg in Part B.
Drug: GSK2838232 IR1 — GSK2838232 will be available as film-coated tablet for oral use
  Arms: GSK2838232 PIB+IR1+IR2
Drug: GSK2838232 IR2 — GSK2838232 will be available as film-coated tablet for oral use
  Arms: GSK2838232 PIB+IR1+IR2
Drug: Placebo PIB — Oral suspension of hydromellulose acetate succinate will be supplied as powder-in-bottle for reconstitution.
  Arms: GSK2838232 PIB (20mg/50 mg/100 mg/200 mg)/Placebo; GSK2838232 PIB (50 mg+100 mg+200 mg)+Placebo
Drug: Ritonavir — It is to be purchased by site. It will be white film-coated ovaloid tablets for oral administration.

SUMMARY:
GSK2838232 is a Human Immunodeficiency Virus (HIV) maturation inhibitor being developed for the treatment of HIV in combination with other antiretroviral therapy (ART). The primary objectives of this study are to investigate the safety, tolerability, and pharmacokinetics (PK) of single and repeat doses of GSK2838232. This study will be a double-blind, placebo-controlled, single and repeat dose escalation study. This study will be conducted in two Parts: single escalating doses (Part 1A and 1B), and repeated escalating once daily (QD) doses for 11 days (Part 2) of GSK2838232 co-dosed with RTV. During Part 1A, single doses of GSK2838232 (as of active pharmaceutical ingredient-powder in bottle [API PiB]) 50 milligrams (mg), 100mg and 200mg will be administered with RTV. Part 1B will evaluate the relative bioavailability of single doses of crystalline active pharmaceutical ingredient (API) Immediate Release Tablet (IR) tablets versus API PiB as reference, administered with RTV. In Part 2, multiple doses of GSK2838232 will be co-administered with RTV 100mg QD for 11 days as sequential dose cohorts. Maximum duration of study participation will be approximately 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age: Between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the Investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, and outside the reference range for the population being studied, may be included only if the Investigator in consultation with the Medical Monitor, if required, agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
* A creatinine clearance (CLcr) >80milliliter/minute (mL/min) as determined by Cockcroft-Gault equation CLcr (mL/min) = (140 - age) * weight (Wt) / (72 * serum creatinine [Scr]) (times 0.85 if female) where age is in years, Wt is in kilogram (kg), and Scr is in units of milligram / decilitre (mg/dL);.
* Body weight >= 50.0 kg (110 pounds [lbs.]) for men and >= 45.0kg (99lbs) for women and body mass index (BMI)
* Male or females of non-reproductive potential:

A female subject is eligible to participate if she is not pregnant [as confirmed by a negative serum human chorionic gonadotrophin (hCG) test], not lactating, and of non-reproductive potential which is defined as:

Pre-menopausal females with one of the following: Documented tubal ligation; Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion ; Hysterectomy; Documented Bilateral Oophorectomy Post menopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels)]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until one week after the last dose of study medication.

Vasectomy with documentation of azoospermia, or Male condom plus partner use of one of the contraceptive options following: Contraceptive subdermal implant that meets the standard operating procedure (SOP) effectiveness criteria including a <1% rate of failure per year, as stated in the product label; Intrauterine device or intrauterine system that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label; Oral Contraceptive, either combined or progestogen alone. Injectable progestogen; Contraceptive vaginal ring; Percutaneous contraceptive patches.

These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The Investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

* Capable of giving signed informed consent as described in Study protocol which includes compliance with the requirements and restrictions listed in the consent form and in protocol.

Exclusion Criteria:

* Alanine aminotransferase and bilirubin >1.0* upper limit of normal (ULN).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities.
* Subjects who have asthma or a history of asthma.
* Medical history of cardiac arrhythmias or cardiac disease or a family and personal history of long QT syndrome
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GlaxoSmithKline (GSK) Medical Monitor, the medication will not interfere with the study procedures or compromise subject safety
* History of regular alcohol consumption within 6 months of the study defined as: For US sites: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams (g) of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150mL) of wine or 1.5 ounces (45mL) of 80 proof distilled spirits.
* Regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates their participation
* Presence of hepatitis B surface antigen (HBsAg), or positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* Screening or baseline cardiac troponin I greater than the 99% cut-off (>.045 nanograms/mL by the Dimension Vista Cardiac troponin assay) for a given assay.
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500mL within 56 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Exclusion Criteria for 48-Hour Screening Holter:

Any symptomatic arrhythmia (except isolated extra systoles). Sustained cardiac arrhythmias (such as atrial fibrillation or flutter, supraventricular tachycardia (>=10 consecutive beats), complete heart block).

Non-sustained or sustained ventricular tachycardia (defined as >= 3 consecutive ventricular ectopic beats).

Any conduction abnormality (including but not specific to left or right incomplete or complete bundle branch block, atrioventricular (AV) block [2nd degree or higher], Wolf Parkinson White (WPW) syndrome etc.).

Sinus Pauses > 3 seconds. 300 or more supraventricular ectopic beats in 24 hours. 250 or more ventricular ectopic beats in 24 hours.

* Any clinically significant abnormal echocardiogram finding. Abnormal echocardiogram findings should be discussed with the Medical Monitor prior to enrolment.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination):

Heart rate for Males <45 and >100 beats per minute (bpm), for females <50 and >100bpm PR Interval <120 and >220 millisecond (msec) QRS duration <70 and >120msec QT interval corrected (Fridericia's) >450msec

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Approximately 10 weeks
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Safety as assessed by absolute values and change from Baseline in hematology parameters -Part 1 | Baseline (Day -1) and up to 10 weeks
  Hematology parameters includes platelet count, red blood cells (RBC) count, mean corpuscular volume (MCV), neutrophils, white blood cells (WBC) count (absolute), mean corpuscular hemoglobin (MCH), lymphocytes, reticulocyte count, mean corpuscular hemoglobin concentration (MCHC), monocytes, hemoglobin, eosinophils, hematocrit and basophils. Hematology parameters will be evaluated at Day -2, Day -1, Day 2, Day 4, Day 14 of each visit.
Safety as assessed by absolute values and change from Baseline in hematology parameters - Part 2 | Baseline (Day-1) and up to Day 31 for each cohort.
  Hematology parameters includes platelet count, RBC count, MCV, neutrophils, WBC count (absolute), MCH, lymphocytes, reticulocyte count, MCHC, monocytes, hemoglobin, eosinophils, hematocrit and basophils. Hematology parameters will be evaluated at Day -1, Day 2, Day 4, day 8, Day 11, Day 14, Day 17, Day 31 for each cohort
Safety as assessed by absolute values and change from Baseline in clinical chemistry parameters -Part 1 | Baseline (Day -1) and up to 10 weeks
  Clinical chemistry parameters includes blood urine nitrogen (BUN), potassium, aspartate aminotransferase (AST), Lipase, Creatinine, Sodium, alanine aminotransferase (ALT), total protein, glucose, chloride, alkaline phosphatase, albumin, magnesium, total carbon dioxide (CO2), total and direct bilirubin, uric acid, calcium, phosphorus and gamma-glutamyl transferase (GGT). Clinical chemistry parameters will be evaluated at Day -2, Day -1, Day 2, Day 4, Day 14 of each visit.
Safety as assessed by absolute values and change from Baseline in clinical chemistry parameters- Part 2 | Baseline (Day-1) and up to Day 31 for each cohort.
  Clinical chemistry parameters includes BUN, potassium, AST, lipase, creatinine, sodium, ALT, total protein, glucose, chloride, alkaline phosphatase, albumin, magnesium, total CO2, total and direct bilirubin, uric acid, calcium, phosphorus and GGT. Clinical chemistry parameters will be evaluated at Day -1, Day 2, Day 4, day 8, Day 11, Day 14, Day 17, Day 31 for each cohort
Safety as assessed by absolute values and change from Baseline in urinalysis parameters-Part 1 | Baseline (Day -1) and up to 10 weeks
  Urinalysis parameters includes specific gravity, pH, glucose, protein, blood and ketones by dipstick, microscopic examination. Urinalysis parameters will be evaluated at Day -2, Day -1, Day 2, Day 4, Day 14 of each visit.
Safety as assessed by absolute values and change from Baseline in urinalysis parameters-Part 2 | Baseline (Day-1) and up to Day 31 for each cohort.
  Urinalysis parameters includes specific gravity, pH, glucose, protein, blood and ketones by dipstick, microscopic examination. Urinalysis parameters will be evaluated at Day -1, Day 2, Day 4, Day 11, Day 14, Day 17, Day 31 for each cohort
Safety as assessed by Blood pressure-Part 1 | 10 weeks
  Systolic and diastolic blood pressure will be measured on Day 1, pre-dose (triplicate) and 1, 2, 4, 6, 8, 12, 24, 48, and 72hr post-dose during each visit.
Safety as assessed by Heart rate -Part 1 | 10 weeks
  Heart rate will be measured on Day 1, pre-dose (triplicate) and 1, 2, 4, 6, 8, 12, 24, 48, and 72hr post-dose during each visit.
Safety as assessed by Blood pressure-Part 2 | 31 days in each cohort
  Systolic and diastolic blood pressure will be measured on Day -1, Day 1 at pre dose (triplicate), and 1hr, 4hr, 24hr, 48hr and 72hr post dose, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11 at pre dose (triplicate), and 1hr, 4hr, 24hr, 48hr and 72hr post dose and at follow up during each cohort.
Safety as assessed by Heart rate -Part 2 | 31 days in each cohort
  Heart rate will be measured on Day -1, Day 1 at pre dose (triplicate), and 1hr, 4hr, 24hr, 48hr and 72hr post dose, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11 at pre dose (triplicate), and 1hr, 4hr, 24hr, 48hr and 72hr post dose and at follow up during each cohort.
Safety as assessed by Electrocardiogram (ECG) parameters-Part 1 | Up to 10 weeks
  12-lead ECG will be conducted pre-dose on Day 1 (triplicate), and 1, 2, 4, 6, 8, 12, 24, 48 72 hour post dose.
Safety as assessed by ECG parameters-Part 2 | 31 days in for each cohort
  A single 12-Lead ECG will be conducted at screening and Day -1, Day 1 at pre dose (triplicate), and 1 hour, 12 hour, 24hour, 48 hour and 72 hour post dose, Day 5, Day 8 and Day 11 at pre dose (triplicate), and 1 hr, 12 hour, 24 hour, 48 hour, and 72 hour post dose and at follow up during each cohort.
Area under the concentration-time curve from time zero (pre-dose) to 24 hours (AUC[0-24]), Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC [0-inf]) in Part 1 | Plasma samples will be collected pre-dose (within 15 minutes prior to dosing) and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose at each study visit
Apparent oral clearance (CL/F) for single dose GSK2838232 in Part 1A | Plasma samples will be collected pre-dose (within 15 minutes [min]prior to dosing) and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose at each study visit during Part 1A.
Area under the concentration-time curve over the dosing interval (AUC[0 tau]) for repeated dose GSK2838232 in Part 2 | Day 1; pre-dose (within 15 min prior to dosing) and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12 and 24 hr post dose.On Day 11; pre-dose (within 15 min prior to dosing) and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hr post dose
Apparent oral clearance (CL/F) for repeated dose GSK2838232 in Part 2 | Plasma samples will be collected on Day 11; pre-dose (within 15 minutes prior to dosing) and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours post dose.
Tmax for repeated dose GSK2838232 in Part 2 | Day 1; pre-dose (within 15 min prior to dosing) and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12 and 24 hr post dose. On Day 11; pre-dose (within 15 min prior to dosing) and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96,120 and 144 hr post dose
Tlag for repeated dose GSK2838232 in Part 2 | Day 1; pre-dose (within 15 min prior to dosing) and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12 and 24 hr post dose. On Day 11; pre-dose (within 15 min prior to dosing) and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96,120 and 144 hr post dose
T1/2 for repeated dose GSK2838232 in Part 2 | Day 1; pre-dose (within 15 min prior to dosing) and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12 and 24 hr post dose. On Day 11; pre-dose (within 15 min prior to dosing) and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96,120 and 144 hr post dose
Tlast for repeated dose GSK2838232 in Part 2 | Day 1; pre-dose (within 15 min prior to dosing) and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12 and 24 hr post dose. On Day 11; pre-dose (within 15 min prior to dosing) and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96,120 and 144 hr post dose
Maximum observed concentration (Cmax) in Part 1 | Plasma samples will be collected pre-dose (within 15 minutes prior to dosing) and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose at each study visit
Concentration at 24 hours post dose (C24) in Part 1 | Plasma samples will be collected pre-dose (within 15 minutes prior to dosing) and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose at each study visit
Last measurable concentration (Clast) in Part 1 | Plasma samples will be collected pre-dose (within 15 minutes prior to dosing) and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose at each study visit
Time of occurence of Cmac (tmax) in Part 1 | Plasma samples will be collected pre-dose (within 15 minutes prior to dosing) and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose at each study visit
Lag time before observation of drug concentrations in sampled matrix (tlag) in Part 1 | Plasma samples will be collected pre-dose (within 15 minutes prior to dosing) and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose at each study visit
Terminal phase half life (t1/2) in Part 1 | Plasma samples will be collected pre-dose (within 15 minutes prior to dosing) and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose at each study visit
Time of last observed quantifiable concentration (t-last) in Part 1 | Plasma samples will be collected pre-dose (within 15 minutes prior to dosing) and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose at each study visit
Cmax of GSK2826232 in Part 2 | Day 1; pre-dose (within 15 min prior to dosing) and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12 and 24 hr post dose.On Day 11; pre-dose (within 15 min prior to dosing) and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hr post dose
Clast of GSK2826232 in Part 2 | Day 1; pre-dose (within 15 min prior to dosing) and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12 and 24 hr post dose.On Day 11; pre-dose (within 15 min prior to dosing) and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hr post dose
Concentration-time curve over the dosing interval (Ctau) of GSK2838232 in Part 2 | Day 1; pre-dose (within 15 min prior to dosing) and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12 and 24 hr post dose.On Day 11; pre-dose (within 15 min prior to dosing) and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hr post dose

SECONDARY OUTCOMES:
AUC (0-inf) in Part 1 | Plasma samples will be collected pre-dose (within 15 minutes prior to dosing) and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose at each study visit
Cmax in Part 1 | Plasma samples will be collected pre-dose (within 15 minutes prior to dosing) and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose at each study visit
AUC(0-tau) in Part 2 | Day 1 pre-dose; 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24 hr post dose. Days 3-10 pre-dose; Day 11; pre-dose and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hr post dose; all pre-dose within 15 min prior to dosing
Cmax in Part 2 | Day 1 pre-dose; 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24 hr post dose. Days 3-10 pre-dose; Day 11; pre-dose and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hr post dose; all pre-dose within 15 min prior to dosing
Ctau in Part 2 | Day 1 pre-dose; 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24 hr post dose. Days 3-10 pre-dose; Day 11; pre-dose and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hr post dose; all pre-dose within 15 min prior to dosing
Pre-dose GSK2838232 plasma concentrations on Day 2-11 in Part 2 | Up to Day 11
Accumulation ratios (Ro) for AUC (0-tau) | Day 1 pre-dose; 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24 hr post dose. Days 3-10 pre-dose; Day 11; pre-dose and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hr post dose; all pre-dose within 15 min prior to dosing
Accumulation ratios (Ro) for Cmax | Day 1 pre-dose; 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24 hr post dose. Days 3-10 pre-dose; Day 11; pre-dose and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hr post dose; all pre-dose within 15 min prior to dosing
Accumulation ratios (Ro) for Ctau (where tau is 24 hours) | Day 1 pre-dose; 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24 hr post dose. Days 3-10 pre-dose; Day 11; pre-dose and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hr post dose; all pre-dose within 15 min prior to dosing

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States